CLINICAL TRIAL: NCT00884364
Title: Exercise During Chemotherapy for Patients With Hematological Malignancies
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Dr. Fernando Dimeo, Dept. of Sports Medicine, Charité Universitätsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: EA4/031/09
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Hematological Diseases; Hematological Malignancies
Keywords: Lymphoma; Leukemia; Multiple myeloma; Hodgkin´s disease; Exercise; Sport; Fatigue; Hematological neoplastic diseases
MeSH Terms: conditions — Hematologic Diseases; Hematologic Neoplasms; Lymphoma; Leukemia; Multiple Myeloma; Hodgkin Disease; Motor Activity; Fatigue | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Behavioral: Fatigue counseling
- Exercise (Experimental)
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise — The patients will carry out an aerobic exercise program consisting of walking on a treadmill for 30 minutes at an intensity of 80% of the maximum heart rate. The training will be carried out three times a week.
  Arms: Exercise
Behavioral: Fatigue counseling — The patients will receive a counseling regarding the causes of fatigue, how to cope with this symptom, and general recommendations about exercise. However, they will not participate at a structured exercise program.
  Arms: Control

SUMMARY:
The trial will evaluate the effects of aerobic exercise in patients undergoing chemotherapy for the treatment of a hematological neoplastic disease.

ELIGIBILITY:
Inclusion Criteria:

* Hematological malignant disease
* Current chemotherapy
* Understanding of written German

Exclusion Criteria:

* Cardiorespiratory, metabolical, osteoarticular or immunological disorders which can be aggravated by exercise
* Pathological stress-ECG at recruitment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-04 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Fatigue | At recruitment and after 12 weeks

SECONDARY OUTCOMES:
Complications | At recruitment and after 12 weeks
Physical performance | At recruitment and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Dimeo, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Section Sports Medicine, Charité Universitätsmedizin Berlin, Hindenburgdamm 30, Berlin, State of Berlin, Germany